CLINICAL TRIAL: NCT05167422
Title: Preliminary Study of a Trusted Messenger Intervention to Promote Vaccine Uptake in Adult Inpatient Psychiatric Hospitals
Brief Title: Trusted Messenger Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey C. Fetter, MD Chief Medical Officer, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 02001055
Record Dates: First submitted 2021-10-05; First posted 2021-12-22 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Vaccine Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Nested quasi-experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trusted Messenger (Experimental): The trusted messenger patient intervention will involve training a small number of staff "trusted messengers" to engage patients informally and assist with building vaccine confidence in brief one- on-one sessions, supported by trusted messengers weekly consultations with a content expert who can answer specific vaccine related questions that patients have over a 3-week period. Trusted messengers will be full time unit employees, selected with the assistance of the nursing supervisor for having excellent rapport with patients (assessed with the Nurse Coordinator Questionnaire) and for having been vaccinated. Mental health workers or nurses may serve in this role. Both inpatient units involved in this study will be grouped into the same vaccination cohort within the hospital, to provide patients in the intervention and the wait list similar opportunities to be vaccinated.
  Interventions: Behavioral: Trusted Messenger
- Standard Care (No Intervention): After a 3-week study period, up to 24 patients on the second unit will receive the trusted messenger intervention and followed for a period of 3 weeks. The trusted messenger intervention will consist of staff who are trained to engage patients informally and assist building social norms for vaccine uptake supported by weekly and as-needed check-ins with a content expert who can answer specific vaccine related questions over a 3 week period.

INTERVENTIONS:
Behavioral: Trusted Messenger — A nested waitlist design in which patients and staff are nested within two inpatient psychiatric units. New Hampshire Hospital staff will be trained to deliver the trusted messenger intervention up to 24 patients on the first unit while the second unit receives care as usual, during which time in-house vaccinations among patients on both units will be tracked in a registry. After a 3-week study period, up to 24 patients on the second unit will receive the trusted messenger intervention and followed for a period of 3 weeks. The trusted messenger intervention will consist of staff who are trained to engage patients informally and assist building social norms for vaccine uptake supported by weekly and as-needed check-ins with a content expert who can answer specific vaccine related questions over a 3 week period.
  Arms: Trusted Messenger

SUMMARY:
The objective of this pilot study is to develop and evaluate test a trusted messenger intervention targeting vaccine hesitancy in patients on an inpatient psychiatric hospital setting with both acute and chronic patients.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give verbal informed consent to participate in the study or able to assent with guardian consent
* Expected to remain in the hospital for the duration of the study
* Mental health diagnosis Demographics
* Male, female, or transgender (no exclusion criteria based on gender or sexual orientation)
* Ages 18 or older
* Any race or ethnicity
* English speaking

Exclusion Criteria:

* Cognitive impairment sufficient to interfere with participant's ability to provide assent
* People who are non-English speakers or who have major visual or hearing impairment will be excluded given the need to converse with the Trusted Messenger verbally
* People who have received any of the available forms of the COVID-19 vaccine, or those with a medical exemption for receiving the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Vaccine acceptance- This will be measured using the COVID Vaccine Hesitancy Questionnaire | Participant is willing to receive the vaccine by the end of week 6 of participation from baseline.
  The participant is willing to receive the COVID-19 vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- New Hampshire Hospital, Concord, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No